CLINICAL TRIAL: NCT04721743
Title: Microbiome as a ThErapeutic Response Biomarker
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled. Investigator left NIH.
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200078; 20-EI-0078
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Uveitis
Keywords: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected Participants: Participants with Uveitis

SUMMARY:
Background:

Uveitis is inflammation inside of the eye. It can cause vision loss. Little is known about the disease. There are few treatment options. Researchers want to learn how the bacteria in the gut might affect how people with uveitis respond to treatment.

Objective:

To investigate the natural bacteria present in the gut and intestines to study whether it might affect uveitis treatment.

Eligibility:

People ages 13 and older with non-infectious uveitis who are enrolled in the ADalimumab Vs. conventional ImmunoSupprEssion for uveitis (ADVISE) trial, and their uveitis is being treated or will be treated with an oral corticosteroid, conventional immunosuppressive drugs, or adalimumab.

Design:

Participants will have 2 study visits at their respective clinical sites. The visits will be 6 months apart. The visits will align with the main ADVISE trial visits.

Participants will give blood samples. A needle will be used to take blood from an arm vein. They will also give stool samples. They will get stool collection kits. They will collect each sample at home and send it to the NIH.

Participants will complete online diet history questionnaires. They will get an ID and password to access the questionnaires. The ID is a unique code. This means it does not contain any personal identifiers. They can complete the questionnaires at home.

Participation in this study will last for 6 months.

DETAILED DESCRIPTION:
Objective: To investigate the potential of gut microbiota as a biomarker of responsiveness to treatment and to evaluate treatment related changes in fecal microbiota composition among posterior segment uveitis patients.

Study Population: Up to 150 participants with uveitis may be enrolled in this study across up to 21 participating sites.

Design: This is a prospective, case-control ancillary study. Participants will be asked to provide a stool sample, blood sample, and complete an on-line Diet History Questionnaire (DHQ). The study will last approximately three years, with two years for recruitment and one year for follow-up. Participants must be co-enrolled in the parent ADVISE protocol (NCT 03828019.) in order to be eligible for this study.

Outcome Measures: The primary outcome answers whether there is a gut microbial signature at baseline that can predict therapeutic response among uveitis patients. Additionally, this study will explore whether the gut microbial ecology change differentially in response to conventional immunosuppressives or tumor necrosis factor inhibitors (TNFi) treatment. Secondary outcomes include exploring if there are molecular or immune phenotypic markers of activity or therapeutic response: To identify molecular correlates of disease activity and treatment response through transcriptional profiling (bulk ribonucleic acid (RNA) sequencing of whole blood samples collected in PAXgene tubes or a similar RNA stabilizing tube) and to identify immunophenotypic correlates of activity and treatment response through flow cytometry analysis (using Transfix tubes or a similar direct draw collection tubes used to stabilize venous blood at the point of collection and preserve whole blood specimens for immunophenotyping by flow cytometry.)

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant has uveitis and is being enrolled in ADVISE parent clinical trial (NCT 03828019)
2. Participant is willing to provide fecal and blood samples at predetermined time points (two time points that coincide with the clinical trial related blood draws)
3. Participant willing to fill the online health and dietary (food frequency) questionnaire (DHQIII)

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Current acute diarrhea
2. Current or recent (within one month) infectious gastroenteritis
3. Current or recent use of systemic antibiotics (previous one month)
4. History of partial gastrectomy or bariatric surgery

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be uveitis participants enrolled as an ancillary study to the ADVISE trial.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Gut microbiome measurement | Study duration
  Answers whether there is a gut microbiome signature at baseline that can predict therapeutic response among uveitis patients and explore whether the gut microbial ecology changes differentially in response to conventional immunosuppressives or tumor necrosis factor inhibitors treatment.

SECONDARY OUTCOMES:
Markers | Study duration
  Explore if there are molecular or immune phenotypic markers of activity or therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-EI-0078.html